CLINICAL TRIAL: NCT00376831
Title: The Efficacy of Midazolam & Ketamine Versus Midazolam & Fentanyl for Sedation in Ambulatory Colonoscopies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOR440806CTIL
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Last update posted 2007-08-10 (Estimated); Status verified 2007-08

CONDITIONS: Colonoscopy; Conscious Sedation
Keywords: colonoscopy; conscious sedation; midazolam; ketamine; fentanyl
MeSH Terms: interventions — Midazolam; Fentanyl; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 0 (Active Comparator): fentanyl
  Interventions: Drug: Midazolam, Fentanyl
- 1 (Active Comparator): ketamine
  Interventions: Drug: KETAMINE, MIDAZOLAM

INTERVENTIONS:
Drug: Midazolam, Fentanyl — fentanyl 0.07 mcg/kg + midazolam 0.05 mg/kg if needed adding midazolam up to a total of 0.1 mg/kg
  Arms: 0
Drug: KETAMINE, MIDAZOLAM — Ketamine 0.25 mg/kg + midazolam 0.05 mg/kg if needed adding midazolam up to a total of 0.1 mg/kg
  Arms: 1

SUMMARY:
Providing adequate sedation and analgesia is an integral part of the practice of colonoscopy procedure.

There are various protocols and methods used to prevent discomfort and alleviate pain. Conscious sedation is one of the options recommended by the American Society for Gastrointestinal Endoscopy, although the choice of the exact protocol is left to the physician's discretion.

This study will attempt to recommend a preferred protocol based on a double blind randomized prospective method.

The efficacy of midazolam and ketamine will be compared to the efficacy of midazolam and fentanyl for sedation in ambulatory colonoscopies.

The results will be compiled from objective data and patient and physician interviews.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for elective colonoscopy at the Soroka Medical Center who have signed an informed consent.

Exclusion Criteria:

1. Hypersensitivity to benzodiazepines
2. Hypersensitivity to benzyl alcohol
3. Hypersensitivity to ketamine
4. Hypersensitivity to opiates
5. Pregnancy
6. Uncontrolled hypertension
7. Myocardial infarct in the last 6 months
8. CVA
9. Chronic pulmonary disease
10. Renal failure
11. Chronic liver disease (CHILD B or C)
12. Elevated ICP, cerebral hemorrhage or cranial SOL.
13. Hypovolemic shock
14. Glaucoma
15. Mental illness
16. Drug or alcohol addiction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2007-01; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Recovery time | 24 hours following colonoscopy

SECONDARY OUTCOMES:
Sedative effect | 24 hours following colonoscopy
Patient compliance | 24 hours following colonoscopy
Side effects | 24 hours following colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: pavel krugliak, md. professor, Principal Investigator — Head of the endoscopic unit at Soroka Medical Center Beer Sheva Israel
Locations (1):
- Soroka Medical Center, Beersheba, Israel